CLINICAL TRIAL: NCT03924518
Title: Adjunctive Granisetron Therapy in Patients With Sepsis or Septic Shock：A Single-center, Randomized, Controlled, Single-blind Clinical Trial
Brief Title: Adjunctive Granisetron Therapy in Patients With Sepsis or Septic Shock
Acronym: GRANTISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-ZZJHZX-009
Record Dates: First submitted 2019-04-15; First posted 2019-04-23 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2021-01

CONDITIONS: Sepsis
Keywords: sepsis; septic shock; granisetron
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Granisetron; Saline Solution

STUDY DESIGN:
Intervention Model Description: The participants in treatment group receive intravenous granisetron. The participants in control group receive normal saline.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- granisetron group (Experimental): 3ml granisetron（3mg） will be diluted in 22 mL of 0.9% normal saline,and the granisetron diluted will be intravenously injected for at 10 minutes， every 8 hours for 4 days or until leaving the ICU(death or transfer from ICU to general ward or discharge), whichever come first.
  Interventions: Drug: Granisetron Hydrochloride
- placebo group (Placebo Comparator): Normal saline 25ml every 8h for 4 days or until leaving the ICU(death or transfer from ICU to general ward or discharge), whichever come first.
  Interventions: Drug: Placebo（Normal saline）

INTERVENTIONS:
Drug: Granisetron Hydrochloride — Granisetron will be diluted with 0.9% saline to ensure that the therapeutic drug and placebo are identical in appearance, and 50 ml syringes will serve as the containers for all intravenous drugs.
  Other Names: Selective 5-hydroxytryptamine 3 receptor inhibitor
  Arms: granisetron group
Drug: Placebo（Normal saline） — therapeutic drug and placebo are identical in appearance, and 50 ml syringes will serve as the containers for all intravenous drugs.
  Other Names: 0.9% saline
  Arms: placebo group

SUMMARY:
In this prospective, single-center,randomized,controlled,single-blind clinical trial,Patients will be randomly assigned to receive granisetron or placebo for 4 days or until leaving the ICU(death or transfer from ICU to general ward or discharge). The primary outcome is all-cause death rate at 28 days.

DETAILED DESCRIPTION:
Investigational drug：Granisetron hydrochloride for injection

Study title：Adjunctive Granisetron Therapy in Patients with Sepsis or Septic Shock:A Single-center,Randomized,Controlled,Single-blind Clinical trial.

Principal Investigator：Professor Ping Chang ,Professor Zhanguo Liu, professor Peng Chen,Department of Critical Care Unit, Zhujiang Hospital, Southern Medical University

Study subjects：Adult septic/septic shock patients with procalcitonin(PCT≥2ng/ml when entering the ICU.

Study phase： Investigator Initiated Trial(IIT)

Study objectives：The objective of the study is to determine whether granisetron, compared to placebo, improve the prognosis of sepsis or septic shock,including the reduction in mortality, the protection of organ function and reduction of inflammatory response,and to determine the safety of granisetron in patients with sepsis.

Study design：A Single-center,Randomized,Controlled,Single-blind Clinical trial.

Medication method： Granisetron treatment group： Follow the guidelines for sepsis in 2016 and recommend routine treatment + 3mg granisetron in 22 ml normal saline every 8 h for 4 days or until leaving the ICU(death or transfer from ICU to general ward or discharge), whichever come first.

Placebo control group：Follow the guidelines for sepsis in 2016 and recommend routine treatment + 25ml normal saline every 8 h for 4 days or until leaving the ICU(death or transfer from ICU to general ward or discharge), whichever come first.

Course：4days

Sample size：154.

Sites：1

Primary endpoint：all-cause death at 28 days

Secondary endpoints:

1. The state of liver function: the serum level of transaminase(AST、ALT)、total bilirubin、direct bilirubin at 1,2,3,4,5 days after randomization
2. The state of lung function:oxygenation index(PaO2/FiO2) at 1,2,3,4,5 days after randomization (the patients treated with extracorporeal membrane oxygenation will not collect this indicator).
3. The state of kidney function:serum level of Creatinine (Cr)、blood urea nitrogen(BUN)、Cystatin(Cys) at 1,2,3,4,5 days after randomization
4. The state of inflammatory response:the serum level of interleukin-6(IL-6) 、C-reactive protein 、Superoxide dismutase(SOD) and erythrocyte sedimentation rate(ESR) at 1,3,5 days after randomization.
5. The state of circulation system: the serum level of lactic acid at 1,2,3,4,5 days after randomization
6. The state of immune function:the serum level of white blood cell(WBC)、lymphocyte at 1, 3, 5 days after randomization,the serum level of cluster of differentiation 4 Tcell(CD4+ Tcell) and cluster of differentiation 8 Tcell(CD8+ Tcell) at 1,5days after randomization.
7. The level of plasma 5-hydroxytryptamine(5-HT) at 1,5 days after randomization.
8. Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score at 1, 3, 5 after randomization
9. Incidence and duration of supportive care for organ dysfunction including vasoactive agents, mechanical ventilation, continuous renal replacement therapy(CRRT)、daily condition of fuid balance
10. The length of stay in ICU

Safety endpoints：

1. adverse events
2. Serious adverse events

ELIGIBILITY:
Inclusion Criteria(Only patients who fully meet the following criteria are eligible to participate in the trial):

* Meets the diagnostic criteria for sepsis-3 developed by the American Society of Critical Care Medicine (SCCM)/European Critical Care Medicine Association (ESICM)
* Age ≥18 years old and age ≤80years old.
* Procalcitonin ≥2ng/ml

Exclusion Criteria:

* Age<18 years, or age>80 years.
* Pregnancy or lactating
* A solid-organ or bone marrow transplant patients.
* Patients with myocardial infarction within the past 3 months.
* Advanced pulmonary fibrosis .
* Patients with cardiopulmonary resuscitation before enrollment.
* HIV-positive patients.
* granulocyte-deficient patients.
* blood/lymphatic system tumors are not remission.
* patients with limited care (lack of commitment to full，aggressive life support).
* patients with long-term use of immunosuppressive drugs or with immunodeficiency.
* patients with advanced tumors.
* patients combined with non-infectious factors leading to the death(uncontrollable major bleeding, brain hernia, etc.).
* surgically unresolved infection sources(such as some intraperitoneal infection etc.)
* patients allergic to granisetron.
* patients with intestinal obstruction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
all-cause mortality rate | 28 days
  All-cause mortality rate from the enrollment to the 28th days

SECONDARY OUTCOMES:
liver function(1) | Day at 1,2,3,4,5 after randomization
  the serum level of Alanine transaminase(ALT)
liver function(2) | Day at 1,2,3,4,5 after randomization
  the serum level of Aspartate transaminase (AST)
liver function(3) | Day at 1,2,3,4,5 after randomization
  the serum level of total bilirubin
liver function(4) | Day at 1,2,3,4,5 after randomization
  the serum level of direct bilirubin
lung function | Day at 1,2,3,4,5 after randomization
  oxygenation index(PaO2/FiO2)，the patients treated with extracorporeal membrane oxygenation will not collect this indicator
kidney function(1) | Day at 1,2,3,4,5 after randomization
  serum level of Creatinine (Cr)
kidney function(2) | Day at 1,2,3,4,5 after randomization
  serum level of blood urea nitrogen(BUN)
kidney function(3) | Day at 1,2,3,4,5 after randomization
  serum level of Cystatin(Cys)
inflammatory response(1) | Day at 1,3,5 after randomization.
  the serum level of interleukin-6(IL-6)
inflammatory response(2） | Day at 1,3,5 after randomization.
  the serum level of C-reactive protein(CRP)
inflammatory response(3） | Day at 1,3,5 after randomization.
  the serum level of superoxide dismutase(SOD)
inflammatory response(4） | Day at 1,3,5 after randomization.
  the serum level of erythrocyte sedimentation rate(ESR)
The level of lactic acid | Day at 1,2,3,4,5 after randomization
  the serum level of lactic acid
immune function(1) | Day at 1, 3, 5 after randomization for test the the serum level of white blood cell(WBC).
  the serum level of white blood cell(WBC)
immune function(2) | Day at 1, 3, 5 after randomization for test the the serum level of lymphocyte.
  the serum level of lymphocyte
immune function(3) | Day at 1,5 after randomization for test the the serum level of CD4+ Tcell.
  the serum level of CD4+ Tcell
immune function(4) | Day at 1, 5 after randomization for test the the serum level of CD8+Tcell.
  the serum level of CD8+Tcell
The level of 5-hydroxytryptamine (5-HT) | Day at 1,5 after randomization.
  The level of plasma 5-HT
Sequential Organ Failure Assessment (SOFA) score | Day at 1, 3, 5 after randomization
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score.SOFA score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.The highest score for each of the six items is 4 points, and the lowest score is 0 points.Finally, the scores of the six items are summed to get the value of the sofa score.The range of the sofa score is 0-24.Higher values represent a worse outcome.
The proportion of patients receiving mechanical ventilation | 28 days
  The proportion of patients receiving mechanical ventilation within 28 days after randomization
The proportion of patients receiving vasoactive drugs | 28 days
  The proportion of patients receiving vasoactive drugs within 28 days after randomization
The proportion of patients receiving renal replacement therapy(CRRT) | 28 days
  The proportion of patients receiving CRRT within 28 days after randomization
The duration of mechanical ventilation | 28 days
  The the duration of mechanical ventilation therapy in hours( This outcome measure is intended only for patients receiving mechanical ventilation)
The duration of vasoactive drugs | 28 days
  The the duration of vasoactive drugs therapy in hours( This outcome measure is intended only for patients receiving vasoactive drugs)
The duration of CRRT | 28 days
  The the duration of CRRT therapy in hours( This outcome measure is intended only for patients receiving CRRT)
ICU length of stay | 28 days
  ICU length of stay

OTHER OUTCOMES:
Incidence of adverse events | 28 days
  A adverse event refers to any adverse medical event that occur after the intervention of trial. The adverse events are not necessarily causally related to the trial treatment.
Incidence of serious adverse events | 28 days
  Any adverse medical event occurs at any dose that meets one or more of the following criteria: 1. causes death 2. life-threatening 3. requires hospitalization or hospitalization for an extended period of time 4. causes permanent or significant disability and functional defects 5. causes deformity

CONTACTS AND LOCATIONS:
Overall Officials: ping Chang, M.D.PhD, Principal Investigator — Department of Critical Care Medicine of Zhujiang Hospital
Locations (1):
- Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
since some data may involve patients privacy ，we have no plans to share data so far，and some data may be shared later depending on the patient's wishes.

REFERENCES:
- [Background] Gong S, Yan Z, Liu Z, Niu M, Fang H, Li N, Huang C, Li L, Chen G, Luo H, Chen X, Zhou H, Hu J, Yang W, Huang Q, Schnabl B, Chang P, Billiar TR, Jiang Y, Chen P. Intestinal Microbiota Mediates the Susceptibility to Polymicrobial Sepsis-Induced Liver Injury by Granisetron Generation in Mice. Hepatology. 2019 Apr;69(4):1751-1767. doi: 10.1002/hep.30361. Epub 2019 Mar 5. PMID 30506577
- [Derived] Guan J, Guo Y, Chang P, Gan J, Zhou J, Wang H, Cen Z, Tang Y, Liu Z, Chen P. Adjunctive granisetron therapy in patients with sepsis or septic shock (GRANTISS): Study protocol for a randomized controlled trial. Medicine (Baltimore). 2019 Sep;98(39):e17354. doi: 10.1097/MD.0000000000017354. PMID 31574878
- See also: Our previous research — https://doi.org/10.1002/hep.30361